CLINICAL TRIAL: NCT02964858
Title: Radiation Dose Optimization in Diffuse Large B- Cell Lymphoma (DOBL) - A Randomised Phase III Non- Inferiority Trial.
Brief Title: Radiation Dose Optimization in Diffuse Large B- Cell Lymphoma.
Acronym: DOBL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Jayant Sastri Goda, Associate Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project No-1627
Record Dates: First submitted 2016-11-12; First posted 2016-11-16 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: NonHodgkin Lymphoma
Keywords: Radiation Dose; Optimization; NHL; DLBCL; R-CHOP
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Arm (Active Comparator): 45 Gy in 25 fractions of 1.8 Gy per fraction over 5 weeks Involved Field radiotherapy (IFRT)/ Involved Site Radiotherapy (ISRT)
  Interventions: Radiation: Standard Arm
- Experimental Arm (Experimental): 36 Gy in 20 fractions of 1.8 Gy per fraction over 4 weeks Involved Field radiotherapy (IFRT)/ Involved Site Radiotherapy (ISRT)
  Interventions: Radiation: Experimental Arm

INTERVENTIONS:
Radiation: Standard Arm — Radiation will be started within 3-4 weeks of completion of chemotherapy. Computed Tomography (CT)scan will be acquired for treatment planning, which will be done using External Beam Planning System. The target volumes will be defined by clinical examination, staging Positron Emission Tomography with CT (PET-CT) and response PET-CT. The staging PET-CT will be fused and co-registered with the planning CT scans for target volume delineation. For Involved Field Radiotherapy,Clinical target volume (CTV) will include the entire nodal region depending on the site involved. For Involved Site RT , CTV will include the involved nodal volume in the staging PET-CT. For extranodal sites, the CTV will include the involved extranodal region as per the staging PET-CT. The total dose will be prescribed to the Planning Target Volume based on dose uniformity guidelines. All patients will be treated with 3 Dimensional Conformal Radiotherapy or Intensity Modulated Radiotherapy where indicated.
  Arms: Standard Arm
Radiation: Experimental Arm — Radiation will be started within 3-4 weeks of completion of chemotherapy. Computed Tomography (CT)scan will be acquired for treatment planning, which will be done using External Beam Planning System. The target volumes will be defined by clinical examination, staging Positron Emission Tomography with CT (PET-CT) and response PET-CT. The staging PET-CT will be fused and co-registered with the planning CT scans for target volume delineation. For Involved Field Radiotherapy,Clinical target volume (CTV) will include the entire nodal region depending on the site involved. For Involved Site RT,CTV will include the involved nodal volume in the staging PET-CT. For extranodal sites, the CTV will include the involved extranodal region as per the staging PET-CT. The total dose will be prescribed to the Planning Target Volume based on dose uniformity guidelines. All patients will be treated with 3 Dimensional Conformal Radiotherapy or Intensity Modulated Radiotherapy where indicated.
  Arms: Experimental Arm

SUMMARY:
The purpose of this study is to compare standard dose radiation of 45 Gray(Gy) in 25 fractions in Non Hodgkin's Lymphoma- Diffuse Large B cell Lymphoma (NHL-DLBCL) to that of 36 Gy in 20 fractions.

The role of radiation in NHL-DLBCL has been addressed in large cooperative trials showing improvement in overall survival and progression free survival with combined modality treatment. The doses of radiation used in these trials are heterogeneous ranging from 30-55 Gray(Gy). There is uncertainty about the optimal dose of radiation needed in aggressive lymphomas. A dose response phenomenon is known in Non- Hodgkin's Lymphoma. Late effects of higher dose radiation in the form of higher risk of stroke, myocardial infarction, thyroid abnormalities and secondary breast cancer are being increasingly identified. Hence it is essential to optimize the dose of radiotherapy for lower toxicity without compromising on efficacy.

DETAILED DESCRIPTION:
Patients who fit the eligibility criteria will be screened for the trial. Patients who consent to participate in the trial will be registered into the trial prior to the start of chemotherapy.

Patient registration / randomization procedure

After completion of staging, the patient is informed about this trial after checking the eligibility checklist.

The patient is informed about this trial, including the following main points: title and aim of the trial, nature of the treatment, side effects, reason for randomization, passing on of data and material samples and the patient's freedom to decide.

The patient receives an information brochure and an informed consent form. The written consent to participate in the trial and to randomization, if needed, in the presence of a witness takes place at least 24 hours after patient briefing. The signed original consent form and the record of the briefing remain in the patient's files. The patient receives a copy of each document. If after completion of staging the patient is qualified for a trial and gives written informed

Consent, then randomization will be performed by statistician at Clinical Research Secretariat, Institutional Review Board. For randomization, the following is required:

* All entry criteria satisfied;
* No exclusion criterion satisfied;
* Staging and stage allocation according to protocol;
* Signed trial consent form in possession of the trial coordinator.

Randomization Patients will be randomized after the completion of 4-6 cycles of chemotherapy just prior to starting radiation.

The stratification variables used are

1. Response: Complete response and partial response.
2. Bulky disease. Bulky is defined as any nodal lesion measuring > 7 cm and mediastinal mass greater than a third of the trans thoracic diameter at any level of thoracic vertebrae as determined by CT and Non bulky is lesion measuring < 7 cm.
3. Revised International Prognostic Index: The negative prognostic factors used for this stratification are age > 60 years, stage III/IV disease, elevated lactate dehydrogenase level, Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2, more than one extranodal site of disease.

I: Very Good Risk: No risk factors. II: Good Risk: 1-2 Risk factors. III: Poor Risk: 3-5 Risk factors.

Radiation Therapy Protocol

Patient's positioning:

The patient positioning and immobilization would vary depending on the site being treated. In general patient will be positioned supine with an immobilization device. Orthogonal lasers will be used for patient alignment. Laser marks will be made on the thermoplastic mask will help in setting up the patient during treatment.

Simulation (patient data acquisition) guidelines. A planning CT scan will be acquired to delineate the target volumes namely gross tumor volume (GTV), clinical target volume (CTV), and planning target volume (PTV).

Patients will be positioned in actual treatment position depending on the site (as described above) on flat table couch with fiducials at a stable bony landmark. CT slices with 5mm thickness will be obtained.

PET CT at baseline will be used to guide the delineation of CTV. It will be fused electronically with the CT simulation scan so that original volumes of interest can be displayed on the simulation CT.

PTV will provide margin around the CTV to compensate for variability in daily treatment set-up. It includes the entire CTV plus a minimum 3D margin of 5 mm.

Dose-volume histograms (DVH) will be generated for each site and the plan will be evaluated in consideration of the expected normal tissue complication probability.

Dose computation. External Beam Planning System of Eclipse (Varian Medical Systems, Palo Alto, USA, V 8.6.14) will be used for generating the plans. Convolution algorithm will be used for dose calculation. The PTV will be treated with any combination of coplanar or non-coplanar 3-dimensional conformal fields shaped to deliver the prescribed dose while minimizing dose to the normal tissue OAR. Field arrangements will be determined by 3 D planning to produce the optimal conformal plan in accordance with volume definitions. The treatment plan used for each patient will be based on an analysis of the volumetric dose including DVH analyses of the PTV and critical organ at risk (OAR). Each field is to be treated daily.

The PTV will be outlined in all relevant planes. The dose distribution in form of isodose lines or dose color wash will be shown in all three planes through the beam axes.

Equipment and tools. Megavoltage beams will be used for treating patients. Beam's Eye View techniques will be used to select the beam isocenter and direction to fully encompass the target volume but minimizing the inclusion of the critical organs in order to select the plan that minimizes the dose to normal tissues. Visual displays in the axial planes to objectively candidate plans and Dose-Volume Histograms will also be part of the treatment planning procedures.

Dose prescription. Normalization of the treatment plan will cover 95% of the PTV with the prescription dose. The minimum PTV dose (to a volume of at least 0.03 cc) must not fall below 95% of the prescription dose. The maximum dose within the PTV must not exceed 107% of the prescribed dose. All RT doses will be calculated with inhomogeneity corrections that take into account the density differences within the irradiated volume (i.e., air, lung, soft tissues, and bones).

Dose recording. The following dose parameters will be recorded.

* Prescription point dose.
* Minimum and maximum dose in the PTV and average dose in the PTV.
* Hot spot outside the PTV.
* Dose to organs at risk

Dose homogeneity.

* The dose will be prescribed to the PTV. Heterogeneity acceptable is 95% - 107%.
* The minimal dose to the target volume, identified in the central plane fields dose distribution, will be 42.75 Gray (Gy) (95% of the protocol dose)in control arm and 34.2 Gy in experimental arm.
* The maximal target dose (defined as the greatest dose in target volume which is delivered to an area greater than 2 cm ), identified in the central plane will be ≤ 107% of the prescribed dose.(48.15 Gy in control arm and 38.52 Gy in experimental arm).
* If Intensity Modulated Radiotherapy (IMRT) is contemplated,International commission on Radiation Units (ICRU) 83 guidelines will be followed.

Treatment Verification. Electronic portal images, will be obtained during the course of treatment on the first day of treatment and once a week thereafter and will be compared with the digitally reconstructed images from CT scan.

Chemotherapy protocol All patients will receive 4-6 cycles of Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisolone (R-CHOP) chemotherapy based on the stage of the disease.

Follow-up Protocol:

All patients will be followed up as follows:

* From completion of radiotherapy to 2 years: first visit at 3 months +/- 1 month and then 6 monthly.
* Thereafter, the patient followed up yearly till death. The following investigations should be performed during every visit.
* Clinical examination, weight, performance status, including the common toxicity criteria for adverse events (CTCAE) v4.0 scale for acute reactions and late effects
* Lactate dehydrogenase ( S LDH), thyroid function test (TFT), Complete blood count (CBC), Renal function test( RFT) and liver function test (LFT) when clinically indicated.
* A Fluoro De-oxy glucose positron emission Tomography with computed tomography (FDG-PET-CT) scan at 3 months after treatment is repeated if there was partial response after completion of chemotherapy (with PET positive disease) and in the event clinical suspicion of relapse.
* 1 year post-radiotherapy:Pulmonary function test ( PFT) , 2D Echo and thereafter based on suspicion.

Treatment in case of progression In case of disease progression or relapse, the patient will be treated with salvage chemotherapy according to the hospital policy.

Treatment toxicity assessment Acute and late toxicity will be assessed using the National Cancer Institute-Common Toxicity Criteria (NCI-CTCAE version 4.0) Criteria of evaluation.

The definitions of endpoints used in this trial are :

Relapse: It is defined as the development of a new lesion either in previously treated area, outside the treated area and distant sites or B-symptoms following complete remission (CR) at least 3 months after end of treatment. If the interval is shorter the event is evaluated as a progression.

Toxic effects: These are measures using the CTCAE version 4 Quality of life (see special section on this) Survival: 1) Event Free Survival (EFS): From the time of randomization till relapse or progression or death due to any cause or death due to disease.

2) Overall Survival (OS): From the time of randomization to death due to any cause /death due to disease.

Response rates will be measured using the Revised response criteria for Lymphoma by International Harmonization Project. The response will be measured as Complete response (CR), Partial response (PR), stable disease (SD) and Progressive disease (PD).

Statistical considerations. Statistical design Sample size calculation. The trial is a non-inferiority design. The expected EFS (Event Free Survival) in control arm is 70% at 2 years based on average EFS of patients treated with R-CHOP in trials from US and Group of adult lymphoma research (GELA) . The maximum acceptable non-inferiority margin is 7% with a hazard ratio of 1.3 corresponding to 63% EFS in experimental arm at 2 years.

With a Type I error (α) of 0.05 (1 sided) and power of test 80%, expected duration of recruitment of 4 years, minimal follow up of 2 years and the total number of events needed 369, the sample size is 754 patients (both arms). Considering an attrition rate of 10%, the total sample size is estimated to be 840 patients (420 in each arm).

* One interim analysis is planned for the primary endpoint at 2.5 years when 25% of the likely number of events (92 events) have been observed. Using the O'Brien stopping rule, the boundaries at interim analysis and final analysis are 3.75 and 1.64 respectively.
* Stopping rule criteria: The experimental arm (reduced dose) will be stopped, and switched over to control arm if on interim analysis, more than 25% events occur in the experimental arm.

Analyses will be conducted in agreement with the intention-to-treat principle. Descriptive statistics will be generated for the range of outcome variables, in particular to gauge whether randomization resulted in a balanced distribution of patients characteristics across the experimental conditions. These include the frequency statistics like mean, median and standard deviation.

Definition of end-points

1. Event Free Survival: From the time of randomization till relapse or progression or death due to any cause or death due to disease.
2. Overall Survival: From the time of randomization to death due to any cause /death due to disease.
3. Local Control: From the time of randomization till the disease is controlled at the site of radiation.

The tests to be used for the endpoints are:

1. To estimate event free survival and overall survival, Kaplan Meier curves will be presented for the two arms, with corresponding median EFS and OS, and survival estimates at 2 years with corresponding 90% confidence intervals (CI).
2. Cox proportional hazard analysis will be used for assessing the effect of different variables on the survival specifically the stratification factors. The treatment effect in terms of hazard ratio will be presented corresponding to 90% CI. Decision making will be based on the upper limit of the 90% confidence interval around the HR for EFS. If the upper limit is below 1.34, the lower dose radiotherapy arm will be declared non-inferior to the standard arm. Survival will also be compared between the two arms by log rank test.
3. Local control and response rates will be compared between the two arms by the logistic regression adjusting for stratification factors.

   The proportion of patients achieving CR rates will be compared by logistic regression adjusting for stratification factors.
4. The incidence of toxicity between the arms will be compared by Logistic regression or Chi square test.
5. The quality of life measures between the arms will be compared by using Mann-Whitney test.

As the trial is assessing non-inferiority, interpretation will be based on the boundaries of the confidence intervals.

Interim Analysis An interim analysis will be performed after 2.5 years of recruitment. At this time point, the likely number of observed events would be 25% of the total number of events.

Independent data monitoring committee (IDMC). The Tata Memorial Hospital Ethics Committee has established the Data and Safety Monitoring Sub Committee for monitoring the conduct of the institutional trials. The Committee has 15 members and meets on the first Friday of every month.

The mandate of the Committee is

* Monitor the overall progress of institutional clinical trials and for ensuring adherence to clinical trial and procedural requirements.
* Ensure the safety of participants, validity of data, projected accrual goals is maintained.
* Ensure that eligibility and evaluation criteria are followed, that risks are not excessive.
* Adverse events are appropriately monitored and reported to the appropriate agencies.
* Enhance the quality of the research by providing the investigator with constructive criticism.

Provide regular reports to the Hospital Ethics Committee

Quality of life assessment

Rationale Patients experience consequences of the disease and of the treatment. These are to be surveyed, and causally linked with the relevant therapies where possible. Thus, quality of life is an endpoint - together with toxicity - for the investigation of consequences of disease and its treatment.

The initial status and chronological course of quality of life of long-term survivors are to be surveyed. Thus, correlations with the overall course of disease can be assessed and ideas for specific supportive measures can be developed.

QOL instrument FACT general and FACT Lymphoma: Functional Assessment of Cancer Therapy - General (FACT-G) is a general quality of life instrument intended for use with a variety of chronic illness conditions. It contains 27 items covering four core HRQOL subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7) The FACT-Lym is used to assess health-related quality of life (HRQOL) in patients with various forms of lymphoma. It contains 42 items (questions) covering HRQOL and common lymphoma symptoms and treatment side-effects. The questionnaire begins FACT-G. The FACT-Lym also includes an Additional Concerns sub-scale (15 items), addressing issues typically experienced by lymphoma patients. Some of the issues covered include pain, itching, night sweats, trouble sleeping, fatigue and trouble concentrating. The FACT-Lym also asks patients about their concerns about lumps and swelling, fevers, infections, weight, appetite, emotional stability and treatment. It has been translated in Hindi, Marathi and Bengali.

Timing of Assessment of QOL QOL will be documented at baseline (pre chemotherapy), beginning of radiotherapy, completion of radiotherapy, at 6 months, 1 year and 2 years after completion of RT.

The QOL forms will be given in person by the trial co-coordinator to the patient during treatment and follow up visit. The patient then returns the completed QoL form directly to the co-coordinator. In case the patient fails to come for the stipulated follow up, patient will be contacted over phone and asked to come for follow up. Alternatively the forms will be sent by the trial coordinator directly to the patient at the appropriate examination dates. The patient returns the completed QOL form directly to the trial coordinator.

Statistical considerations Data will be analysed using descriptive statistics, graphical format and longitudinal modeling.

Forms and procedures for collecting data

Consent Form After patient has consented to the trial, a signed informed consent is obtained. It should bear the signatures of the patient as well as the Chief Investigator or co- investigator of the trial.

Case report forms The case report forms will be filled once the patient is screened for the study and has given his or her consent for participation in the study.

Data flow

* All data which is to be collected is documented on standardized case report forms (CRFs) by the treating physician or other person given the responsibility for documentation.
* If an entry has to be corrected, this should be done using a single line to delete this entry. In addition to the correct and valid text, the date of correction and the signature of the correcting physician or authorized documenting person are to be entered.
* In case of missing or inconsistent data, the physician are contacted for further information. Patients are also contacted over phone if they miss to come for regular follow up.

Reporting adverse events In this section, the classification and documentation / reporting of adverse events is described.

Adverse events are to be recorded on the documentation forms for treatment and follow-up. If an adverse event occurs, the SAE form is completed and sent to the trial coordination center: within 24 hours in the case of fatal or life-threatening events.

The regular toxicity examinations before, during and after treatment are done as described before.

Definitions An Adverse Event (AE) is defined as any untoward medical occurrence or experience in a patient or clinical investigation subject which occurs following the administration of the trial medication regardless of the dose or causal relationship. This can include any unfavorable and unintended signs (such as rash or enlarged liver), or symptoms (such as nausea or chest pain), an abnormal laboratory finding (including blood tests, x-rays or scans) or a disease temporarily associated with the use of the protocol treatment.(ICH-GCP).

An Adverse Drug Reaction (ADR) is defined as any response to a medical product, that is noxious and/or unexpected, related to any dose. (ICH-GCP).

Response to a medicinal product (used in the above definition) means that a causal relationship between the medicinal product and the adverse event is at least a reasonable possibility, i.e. the relationship cannot be ruled out.

An Unexpected Adverse Drug Reaction is any adverse reaction for which the nature or severity is not consistent with the applicable product information (e.g., Investigators' Brochure). (ICH-GCP).

A Serious Adverse Event (SAE) is defined as any undesirable experience occurring to a patient, whether or not considered related to the protocol treatment. A Serious Adverse Event (SAE) which is considered related to the protocol treatment is defined as a Serious Adverse Drug Reaction (SADR).

Adverse events and adverse drug reactions which are considered as serious are those which result in:

* death
* a life threatening event (i.e. the patient was at immediate risk of death at the time the reaction was observed)
* hospitalization or prolongation of hospitalization
* persistent or significant disability/incapacity
* any other medically important condition (i.e. important adverse reactions that are not immediately life threatening or do not result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed above.

Reporting procedure Recording of adverse events (including known adverse drug reactions).

* All adverse events and known adverse reactions during radiotherapy are to be evaluated immediately after occurrence and recorded on the regular documentation forms.
* Adverse events and known adverse drug reactions possibly connected with radiotherapy are assessed according to the criteria and recorded on the CRF.
* Adverse events and known late radiation toxicity occurring during follow-up are recorded on the CRF.

Recording of serious adverse events:

All Serious Adverse events will be reported according to the world health organisation (WHO) guidelines .The SAE's will be reported only after the randomization as the study is evaluating the efficacy of the radiation arms.

All serious adverse events (SAE) according to the definition above are to be documented by the treating physician on the SAE-form as well as on the corresponding regular documentation forms.

On the SAE-form, the treating physician must assess the causal relationship (if any) between the SAE and administration of trial medication. Evaluation scale for causal relationship: related/unrelated/ expected/ unexpected.

If the SAE was fatal or life-threatening, the completed SAE form must be sent to Institutional Review Board (IRB) within 24 hours. A detailed medical report must follow every SAE form within 10 further days to the IRB.

Furthermore, all SAEs occurring during the trial which could endanger the safety of participants or the performance of the trial must be reported to the ethics committee.

Finally, the treating physician must report serious adverse events in compliance with professional codes of practice.

Quality assurance Radiation quality Assurance

1. Initiation visit: Explaining to the physicians and physicists about the trial contouring and planning requirements.
2. Credentialism of physicians and physicists involved in the contouring and planning of the cases for first 4-5 cases. To check for adherence to the protocol parameters.
3. Record of all the plans.
4. Systematic chart reviews.

Control of data consistency Data from case record forms can be entered only after a check of completeness and plausibility. Data entry is made by the qualified trial coordinators. Furthermore, data are cross-checked for plausibility with previously entered data for that patient. After the first data entry has been successfully completed, a second data typist repeats the data input and makes corrections where necessary. Retrospective alterations of data are recorded in an audit table.

Ethical considerations Patient protection The responsible investigator will ensure that this study is conducted in agreement with either the Declaration of Helsinki (Tokyo, Venice, Hong Kong, Somerset West and Edinburgh amendments) or the laws and regulations of the country, whichever provides the greatest protection of the patient.

The protocol has been written, and the study will be conducted according to the ICH Harmonized Tripartite Guideline for Good Clinical Practice.The protocol was be approved by the Local Hospital Ethics Committees.

Subject identification Each patient would be assigned a trial number and help in anonymity of the patient.

Informed consent All patients will be informed of the aims of the study, the possible adverse events, the procedures and possible hazards to which he/she will be exposed, and the mechanism of treatment allocation. They will be informed as to the strict confidentiality of their patient data, but that their medical records may be reviewed for trial purposes by authorized individuals other than their treating physician. The patient informed consent statement in English, Hindi and Marathi is being attached as a separate document along with the protocol.

It will be emphasized that the participation is voluntary and that the patient is allowed to refuse further participation in the protocol whenever he/she wants. This will not prejudice the patient's subsequent care. Documented informed consent will be obtained for all patients included in the study before they are registered or randomized in the study. This must be done in accordance with the national and local regulatory requirements.

The informed consent procedure must conform to the ICH guidelines on Good Clinical Practice. This implies that "the written informed consent form should be signed and personally dated by the patient or by the patient's legally acceptable representative".

ELIGIBILITY:
Inclusion Criteria:

* Histological Diagnosis of NHL- DLBCL.
* Eligible for RT after R-CHOP.
* ECOG 0-3.
* 18 - 65 years.
* Stage I-IV.
* Patients should receive at least 4 cycles of R-CHOP chemotherapy.
* Patients with all extranodal disease except the ones mentioned in the exclusion criteria.
* Able to understand and willing to provide informed consent for participation in the trial.

Exclusion Criteria:

* HIV positive status.
* Relapse or progression of disease during chemotherapy.
* Prior history of chemotherapy
* Prior history of radiotherapy.
* Systemic lymphomas with CNS involvement.
* Primary extranodal Testicular Lymphomas.
* Primary extranodal central nervous system (CNS) Lymphomas.
* Primary extranodal Stomach DLBCL
* Primary extranodal Intestinal DLBCL
* Patients >3 extranodal sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-03 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 2 years
  From the time of randomization till relapse or progression or death due to any cause or death due to disease.
  Assessment by physiological parameter

SECONDARY OUTCOMES:
Local Control Rate | 2 years
  From the time of randomization till the disease is controlled at the site of radiation.
  Assessment by physiological parameter.
Overall Survival | 2 years
  From the time of randomization to death due to any cause /death due to disease. assessment by physiological parameter
Overall response rate | 3 months
  Assessment by physiological parameter
Late toxicity | 2 years
  Assessment by physiological parameter
Acute toxicity | During radiation to 6 weeks from the end of radiation
  Assessment by physiological parameter
Quality of Life scores | 2 years
  assessment by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Sastri Goda, M.D, Principal Investigator — Professor,Tata Memorial Centre
Locations (1):
- Tata Memorial Center, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes